CLINICAL TRIAL: NCT06669585
Title: Cannabis Observations on Brain Waves, Retrieval, and Attention: Experiment 3 (COBRA)
Brief Title: Cannabis Observations on Brain Waves, Retrieval, and Attention: Experiment 3
Acronym: COBRA 3
Status: Recruiting | Type: Observational
Sponsor: L. Cinnamon Bidwell (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, L. Cinnamon Bidwell, Associate Professor, University of Colorado, Boulder
Organization: University of Colorado, Boulder (Other)
Other Study IDs: 20-0309: Experiment 3; R01DA052431 (NIH)
Record Dates: First submitted 2024-10-23; First posted 2024-11-01 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-10

CONDITIONS: Cannabis; Memory; Electroencephalography
Keywords: Cannabis; Memory; Electroencephalography
MeSH Terms: conditions — Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples collected for cannabinoid quantification and DNA analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Cannabis (smoked flower) — Self-Directed Use (ad-libitum)

SUMMARY:
This study investigates the impact of ∆9-tetrahydrocannabinol (THC) and cannabidiol (CBD) on recognition memory in healthy, regular cannabis users. Participants complete the same recognition memory task after self-administering one of two different strains of cannabis flower one day and while not intoxicated another day. Event-related potentials (ERPs) are measured via electroencephalogram (EEG) during the recognition memory task. Blood is collected to quantify THC and CBD exposure. Participants also complete self-report measures of medical history, sleep quality, subjective cognitive function, physical activity, psychological functioning, substance use, and acute drug effects.

DETAILED DESCRIPTION:
Previous research has established cannabis's harmful cognitive impact, with particularly robust and consistent effects in the domain of episodic memory. However, prior work has not sufficiently considered that the memory effects of cannabis are the compound action of different cannabinoids, which vary in their pharmacology and effects. Specifically, CBD, a non-psychotomimetic component of cannabis (doesn't produce a "high"), is thought to have cognitively protective properties and may mitigate some of the harmful effects of THC. Further, few prior studies have tested the effects of high potency strains that are commonly available.

This study tests the effects of commercially available cannabis flower strains on recognition memory performance and ERPs that are related to different underlying memory processes in healthy, regular cannabis users. An episodic memory task is used to assess recognition memory, which asks participants to discriminate between previously studied and non-studied items using pictures as stimuli. Participants complete the same memory task while intoxicated one day and not intoxicated another day. A THC-dominant strain and a strain containing both THC and CBD are included in the study. Participants self-administer one of the two cannabis strains prior to memory encoding and retrieval.

Blood is collected to determine THC and CBD exposure, as well as to explore how genetic variation in genes related to cannabinoid metabolism, cannabis-related behavior, and neurocognitive function associate with memory function before and after cannabis use. Participants also complete self-report measures of medical history, sleep quality, subjective cognitive function, physical activity, psychological functioning, substance use, and acute drug effects.

ELIGIBILITY:
Inclusion Criteria:

1. Must be between the ages of 21 and 40 and provide informed consent;
2. Must be right-handed (Laterality Quotient > 60 on Edinburgh Handedness Inventory - Short Form);
3. Must use cannabis at least 4 days during the month;
4. Must be a cannabis user for at least a year;
5. Must self-report not using other illicit recreational drugs (e.g., cocaine, benzodiazepines (non-prescription), opiates (non-prescription), MDMA, sedatives, or methamphetamine) in the past 30 days, during the Pre-Screening;
6. Must not test positive on a urine toxicology test for drugs of abuse at the Baseline appointment;
7. Must not be using psychotropic medications, however anti-depressant, non-benzodiazepine anti-anxiety, and ADHD medications are ok. ADHD medication users must be willing to abstain from ADHD medication use on appointment days;
8. Must not be a regular nicotine user (≤4 days per week; cigarette, E-cigs, or smokeless);
9. Must not have used caffeine or nicotine (cigarette, E-cigs, or smokeless) for 4 hours before each appointment;
10. Must have a breath alcohol level of 0 at Baseline appointment (to sign consent form);
11. Must not be actively seeking or in treatment for any substance use disorder;
12. Female subjects must not be or trying to become pregnant (as indicated by a pregnancy test administered at Baseline appointment);
13. Must not be in treatment for psychotic disorder or bipolar disorder; or have a history with these disorders;
14. Must not have any physical characteristics (e.g., thick hair, head size exceeding the limit of the net, dyed hair) or experience any technical difficulties during testing that result in a poor-quality EEG recording.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Community sample of healthy, regular cannabis users in the Boulder and Denver areas
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Difference in ERP amplitude (FN400) | Intoxicated session and not-intoxicated session (about 1 week)
  Electroencephalography is used to quantify FN400.
Difference in ERP amplitude (parietal) | Intoxicated session and not-intoxicated session (about 1 week).
  Electroencephalography is used to quantify parietal ERP effects.
Difference in retrieval memory accuracy | Intoxicated session and not-intoxicated session (about 1 week)
  Accuracy will be used to assess task performance.
Difference in retrieval memory performance | Intoxicated session and not-intoxicated session (about 1 week)
  Reaction time will be used to assess task performance.

SECONDARY OUTCOMES:
Change in Positive and Negative Affect Schedule (PANAS) | Before and after acute cannabis use during intoxicated session
  The PANAS is Self-report measurement of positive and negative affect. Both subscales range from 1 - 50, with a higher score on the positive affect scale indicating higher positive affect and a higher score on the negative affect scale indicating higher negative affect.
Change in Drug Effects Questionnaire (DEQ) | Before and after acute cannabis use during intoxicated session
  The DEQ is a visual analogue scale of measure of acute drug effects. Participants are asked 5 questions on the DEQ, each of which range from 0 - 100, with higher values for each item indicating greater drug effect.
Change in Addiction Research Center Inventory (ARCI-M) | Before and after acute cannabis use during intoxicated session
  The ARCI-M is a self-report measure of subjective effects of marijuana. This is a 12-item true-false task, in which higher (true) scores indicate greater intoxication.
Change in Marijuana Craving Questionnaire | Before and after acute cannabis use during intoxicated session
  The Marijuana Craving Questionnaire is a self-report measure of marijuana craving. Participants complete 8 questions ranging from 0 - 10, with a higher score indicating greater cannabis craving and somatic symptoms.
Change in Profile of Mood States (POMS) | Before and after acute cannabis use during intoxicated session
  The POMS is a self-report measure of mood. Participants complete 27 mood-related items ranging from 0 - 4, with higher scores indicating greater levels of specific mood states.
Change in Alcohol Craving Questionnaire | Before and after acute cannabis use during intoxicated session
  The Alcohol Craving Questionnaire is a self-report measure of alcohol craving. This is a 2-item scale with each item ranging 0 - 10, with higher scores indicating greater alcohol craving.
Change in State Adapted Paranoia Checklist-Brief (SAPC-B) | Before and after acute cannabis use during intoxicated session
  The SAPC-B is a self-report measure of paranoia. Participants complete 5 items each ranging from 0 - 10, with higher scores indicating greater feelings of paranoia.
Difference in circulating cannabinoid concentration | Baseline, intoxicated session, and not-intoxicated session (about 3 weeks total over all three sessions)
  Blood levels of THC and CBD will be quantified.

OTHER OUTCOMES:
Exploratory: Correlations between genes related to cannabinoid metabolism, cannabis-related behavior, and neurocognitive function with ERPs and recognition memory performance | Baseline, intoxicated session, and not-intoxicated session (about 3 weeks total over all three sessions)
  DNA samples are collected from a baseline blood sample.
Exploratory: Moderation of primary effects by baseline sleep quality using the Patient-Reported Outcomes Measurement Information Systems (PROMIS) | Baseline, intoxicated session, and not-intoxicated session (about 3 weeks total over all three sessions)
  This is a baseline measure of participant sleep disturbance. Participants complete 4 items, for a total scale score from 4 - 20, with higher scores indicating more sleep disturbance.
Exploratory: Moderation of primary effects by baseline affective symptoms using the Depression Anxiety Stress Scale (DASS) | Baseline, intoxicated session, and not-intoxicated session (about 3 weeks total over all three sessions)
  This is a baseline measure of affective symptoms. Participants complete three separate subscales assessing depression, anxiety, and stress, each with 7 items and with higher scores indicating greater levels of depression, anxiety, and stress.
Exploratory: Moderation of primary effects by baseline substance use history using the Timeline Followback (TLFB) | Baseline, intoxicated session, and not-intoxicated session (about 3 weeks total over all three sessions)
  This is a baseline measure of substance use history. Participants report their substance use over the last 30 days prior to the baseline appointment.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Curran, PhD, Principal Investigator — University of Colorado, Boulder
Locations (1):
- Center for Innovation and Creativity (CINC), Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CUChange Study Website — https://www.colorado.edu/center/cuchange/cobra-0